CLINICAL TRIAL: NCT06920862
Title: Effectiveness of Multi-Modal Digital Interventions for Adolescent Weight Management: A Randomized Controlled Trial
Brief Title: Multi-Modal Digital Interventions for Adolescent Weight Management
Acronym: M2DI-AWM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Pei-Ching Liu, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTYMCTU
Record Dates: First submitted 2025-03-12; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Adolescent; Weight Change, Body; Weight Stigma
MeSH Terms: conditions — Pediatric Obesity; Body Weight Changes; Weight Prejudice

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Modal Digital Intervention Group (Experimental): Participants in this group will receive a multi-modal digital intervention designed to enhance healthy weight control behaviors among overweight and obese adolescents.
  1. Intervention Components: The intervention integrates AI-driven coaching, interactive platforms, gamified applications, and real-time feedback mechanisms.
  2. Session Structure: Participants will complete biweekly intervention sessions (2 hours each) over a 3-month period.
  3. Theoretical Framework: The intervention is grounded in the Theory of Planned Behavior (TPB) to target attitudes, subjective norms, and perceived behavioral control regarding weight control behaviors.
  4. Digital Platform: Participants will have access to the Virti platform, where they will receive personalized guidance and feedback.
  Interventions: Behavioral: Multi-Modal Digital Intervention
- Control Group (General Health Education) (Active Comparator): General Health Education sessions covering basic principles of nutrition, physical activity, and lifestyle modifications for weight management. These sessions will be delivered using traditional educational methods (e.g., brochures, videos, lectures).
  Interventions: Behavioral: Multi-Modal Digital Intervention

INTERVENTIONS:
Behavioral: Multi-Modal Digital Intervention — Participants in this group will receive a multi-modal digital intervention designed to enhance healthy weight control behaviors among overweight and obese adolescents.
  1. The intervention integrates AI-driven coaching, interactive platforms, gamified applications, and real-time feedback mechanisms.
  2. Participants will complete biweekly intervention sessions (2 hours each) over a 3-month period.
  3. The intervention is grounded in the Theory of Planned Behavior (TPB) to target attitudes, subjective norms, and perceived behavioral control regarding weight control behaviors.
  4. Participants will have access to the Virti platform, where they will receive personalized guidance and feedback.

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of a multi-modal digital intervention, based on the Theory of Planned Behavior (TPB), in promoting healthy weight control behaviors among overweight and obese adolescents. This study also aims to reduce the risk of unhealthy weight control behaviors by leveraging artificial intelligence-driven coaching, interactive platforms, gamified applications, and real-time feedback mechanisms.

The main questions this study aims to answer are:

1. Can a multi-modal digital intervention effectively modify adolescents' primary beliefs underlying TPB constructs (attitude, subjective norms, and perceived behavioral control)?
2. How do TPB constructs influence weight control intentions, and how do these intentions translate into either healthy or unhealthy weight control behaviors? What role do adolescents' body image, body satisfaction, and mental health play in moderating the relationship between weight control intention and behavior?

Participants will:

1. Be adolescents aged 12-18 years with a BMI ≥ 85th percentile.
2. Be randomly assigned to either the intervention group (multi-modal digital intervention) or the control group (general health education).
3. Engage in AI-driven coaching, interactive digital sessions, and gamified experiences tailored to TPB constructs.
4. Complete biweekly sessions over a period of three months (each session lasting two hours).
5. Receive personalized feedback and real-time monitoring through the Virti platform.
6. Participate in follow-up assessments at one month and three months post-intervention.

Researchers will compare the intervention group to the control group to determine whether the multi-modal digital intervention leads to a higher adoption of healthy weight control behaviors and a lower prevalence of unhealthy weight control behaviors.

DETAILED DESCRIPTION:
Adolescent obesity remains a global public health challenge with far-reaching implications for physical and psychological well-being. In Taiwan, the prevalence of overweight and obesity among adolescents aged 13-18 has exceeded 30%, mirroring trends observed worldwide. The COVID-19 pandemic has further exacerbated this issue, intensifying weight gain among youth due to disrupted routines, reduced physical activity, poor sleep hygiene, and increased consumption of energy-dense foods. Despite growing awareness and reported intentions to manage weight among adolescents, there remains a substantial gap between intention and sustained healthy behavior.

This study seeks to bridge this intention-behavior gap through the development and evaluation of a multi-modal digital intervention, grounded in the Theory of Planned Behavior (TPB). TPB posits that intention-the most proximal predictor of behavior-is influenced by three constructs: attitude, subjective norm, and perceived behavioral control. Each construct is shaped by a distinct set of beliefs, including behavioral, normative, and control beliefs. However, limited research has explored how these constructs interact to promote healthy weight control behaviors or inadvertently contribute to unhealthy practices such as meal skipping, purging, or misuse of diet pills.

Building on the PI's previous qualitative and quantitative studies validating TPB in Taiwanese adolescents with obesity, this project designs an intervention that targets these belief systems directly. The intervention integrates artificial intelligence-driven virtual coaching, virtual reality (VR)-based simulation scenarios, gamified applications, and real-time feedback and monitoring through the Virti digital platform. Each intervention module is specifically aligned with a TPB construct:

Module A (Attitude): Uses persuasive VR messages to emphasize benefits of healthy weight control (e.g., appearance, health improvement).

Module B (Subjective Norm): Reinforces perceived social support through peer modeling and family involvement.

Module C (Perceived Behavioral Control): Builds self-efficacy by offering coping strategies to overcome common barriers (e.g., dealing with food sharing, time constraints).

The intervention will be delivered biweekly over three months, with each session lasting approximately two hours. Participants will interact with the virtual nurse avatar, respond to scenario-based questions, and receive personalized feedback. Data collection will occur at baseline, one month, and three months post-intervention.

The randomized controlled trial will enroll adolescents aged 12-18 years with a BMI at or above the 85th percentile, recruited from junior and senior high schools in Taipei. Stratified randomization will ensure balanced group assignment across districts. The intervention group will receive the full TPB-based digital program, while the control group will receive standard health education.

To evaluate intervention efficacy, the study will utilize:

TPB-based questionnaires measuring belief constructs and intention,

A weight control behavior scale distinguishing healthy vs. unhealthy practices,

Standardized tools to assess body image (MBSRQ) and mental health (PHQ-A),

Anthropometric and body composition measurements.

Quantitative data will be analyzed using mixed-design ANOVA and structural equation modeling (SEM) to assess changes over time and the mediating role of psychological factors. Thematic analysis of qualitative data (collected via platform interaction and interviews) will further elucidate adolescents' experiences and the intervention's impact.

This research is expected to make a significant contribution by:

Unpacking the cognitive mechanisms that translate weight control intentions into specific behaviors,

Demonstrating how digital interventions can be effectively tailored using TPB constructs,

Offering an innovative, scalable, and theory-driven model for adolescent obesity intervention that prioritizes psychological safety, personalization, and user engagement.

Ultimately, this study aims to inform policy and practice by providing empirical evidence for the use of AI-enhanced, VR-integrated interventions to promote healthy lifestyle behaviors among adolescents-a critical population for early preventive efforts.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years.
* Body Mass Index (BMI) ≥ 85th percentile according to the Health Promotion Administration (HPA) standards.
* Willing to participate in a digital intervention for weight control.
* At least one parent or guardian provides consent for participation.
* Able to understand and use digital devices (smartphones, tablets, or computers).

Exclusion Criteria:

* Significant communication barriers (e.g., severe speech, hearing, or cognitive impairments).
* Psychiatric disorders that affect interpersonal interaction (e.g., schizophrenia, severe depression).
* Previous negative experiences with digital health interventions (VR or AI-based coaching).
* Severe motion sickness that affects the ability to use VR-based tools.
* Currently enrolled in another weight management program that may interfere with study outcomes.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Weight Control Behaviors as Measured by the Weight Control Behavior (WCB) Scale | Baseline (T0), 1 month post-intervention (T1), 3 months post-intervention (T2)
  This outcome measures the change in healthy weight control behaviors among overweight and obese adolescents following the intervention.
  Healthy behaviors include increased physical activity, improved dietary habits (e.g., higher intake of fruits and vegetables), reduced consumption of sugary drinks, and portion control.
  Data will be collected using the healthy subscale of the Weight Control Behavior (WCB) Scale, a validated tool with a score range from 0 to 100.
  Higher scores reflect greater engagement in healthy weight control behaviors. Data will be analyzed as mean change from baseline at T1 and T2.
Change in Unhealthy Weight Control Behaviors as Measured by the Weight Control Behavior (WCB) Scale | Baseline (T0), 1 month post-intervention (T1), and 3 months post-intervention (T2)
  This outcome measures the change in unhealthy weight control behaviors among overweight and obese adolescents following the intervention.
  Unhealthy behaviors include meal skipping, fasting, using diet pills or other weight-loss supplements, and extreme restriction.
  Data will be collected using the unhealthy subscale of the Weight Control Behavior (WCB) Scale, a validated tool with a score range from 0 to 100.
  Higher scores reflect greater frequency of unhealthy behaviors. Data will be analyzed as mean change from baseline at T1 and T2.

SECONDARY OUTCOMES:
Change in TPB Constructs (Attitude, Subjective Norm, and Perceived Behavioral Control) as Measured by the Theory of Planned Behavior (TPB) Questionnaire | Baseline (T0), 1 month (T1), and 3 months (T2) post-intervention
  This outcome measures changes in three key cognitive constructs-attitude, subjective norm, and perceived behavioral control-regarding weight control behaviors among adolescents. These constructs are assessed using a validated Theory of Planned Behavior (TPB) Questionnaire, developed and tested in prior adolescent obesity studies.
  Each construct is measured using multiple items rated on a 7-point Likert scale (ranging from -3 = strongly disagree to +3 = strongly agree). Higher scores indicate more favorable attitudes, stronger perceived social support (subjective norm), and greater confidence in one's ability to perform weight control behaviors (perceived behavioral control).
  Changes will be reported as mean score differences from baseline at T1 and T2 for each construct separately.
Change in Body Mass Index (BMI) | Baseline (T0) and 3 months post-intervention (T2)
  Body Mass Index (BMI) will be calculated using measured weight (kg) and height (m) (BMI = kg/m²). Measurements will be taken using standardized digital scales and stadiometers.
  Changes in BMI will be analyzed as the mean difference from baseline to post-intervention to evaluate changes in body weight status.
Change in Body Fat Mass (kg) as Measured by InBody 770 | Baseline (T0) and 3 months post-intervention (T2)
  This outcome measures changes in total body fat mass (kg) using InBody 770, a validated bioelectrical impedance analysis (BIA) device.
  Fat mass will be reported in kilograms, and changes will be analyzed as mean difference from baseline.
Change in Lean Body Mass (kg) as Measured by InBody 770 | Baseline (T0) and 3 months post-intervention (T2)
  This outcome assesses changes in lean body mass (kg), also measured using the InBody 770 device.
  Lean mass includes muscle and other non-fat tissue. Results will be reported as mean change from baseline.
Change in Body Image as Measured by the Multidimensional Body-Self Relations Questionnaire (MBSRQ) | Baseline (T0) and 3 months post-intervention (T2)
  This outcome assesses changes in body image among adolescents using the MBSRQ, a validated instrument that evaluates multiple dimensions of body-self relations (e.g., appearance evaluation, appearance orientation).
  Scores from relevant subscales will be analyzed as mean score changes from baseline to post-intervention. Higher scores indicate more positive body image and greater satisfaction with one's appearance.
Change in Self-Esteem as Measured by the Multidimensional Body-Self Relations Questionnaire (MBSRQ) | Baseline (T0) and 3 months post-intervention (T2)
  This outcome evaluates changes in self-esteem-related dimensions of body image, particularly self-classified weight and appearance orientation, as assessed by subscales of the MBSRQ.
  Changes will be reported as mean differences in scale scores from baseline to 3 months, where higher scores represent greater self-confidence in body-related self-perception.
Change in Depression Symptoms as Measured by the Patient Health Questionnaire for Adolescents (PHQ-A) | Baseline (T0) and 3 months post-intervention (T2)
  This outcome examines changes in depressive symptoms using the PHQ-A, a 9-item, self-report screening tool adapted from the PHQ-9 for adolescent populations.
  Scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
  The primary analysis will assess mean score change from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
Due to ethical and confidentiality concerns, individual participant data will not be shared.